CLINICAL TRIAL: NCT01867632
Title: Does Acellular Dermal Matrix Reduce Fistula Rate in Primary Palatoplasty
Brief Title: Acellular Dermal Matrix in Primary Palatoplasty
Status: Completed | Type: Observational
Sponsor: Mirko S. Gilardino (Other)
Responsible Party: Sponsor-Investigator, Mirko S. Gilardino, Director, Plastic Surgery Residency Program, Assistant Professor of Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 12-073-PED
Record Dates: First submitted 2013-05-25; First posted 2013-06-04 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Cleft Palate
Keywords: Palatoplasty; Acellular Dermal Matrix
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective group: Prospective cohort where all patients routinely received ADM during cleft palate surgery. A tailored piece of Acellular Dermal Matrix will be placed between the oral and nasal layers at the time of a Furlow Palatoplasty for repair of a Cleft Palate.
  Interventions: Device: Acellular Dermal Matrix
- Retrospective group: Retrospective cohort of cleft palate patients treated at the same institution and by the same surgeon. These patients received ADM selectively for certain cases (tenuous nasal layer closure, tight oral closure, wide cleft).

INTERVENTIONS:
Device: Acellular Dermal Matrix
  Other Names: DermaMatrix
  Groups: Prospective group

SUMMARY:
The goal of the present study is to definitely determine whether the use of acellular dermal matrix (ADM) during primary cleft palate repair decreases the rate of fistula formation. Although individual studies have described promising advantages to its use in cleft palate surgery, no consensus currently exists. Without concrete evidence, one must question the whether the increased cost, time and potential patient risk (human derived tissue) to patients justifies its use in primary cleft palate repair.

DETAILED DESCRIPTION:
There has been a change in the standard practice at the Montreal Children's Hospital where the senior author has shifted from selected application of ADM in certain cases to routine use of ADM in all cleft palate cases. This study is an observational study comparing a prospective cohort group receiving ADM routinely to a retrospective historical cohort group without routine use of ADM.

Objectives of the study:

Primary objectives:

The primary objective of this study is to determine whether routine use of ADM would lower the incidence of palatal fistula in patients undergoing primary cleft palate repair.

Secondary objectives:

1. Incidence of wound dehiscence
2. Incidence of wound infection
3. Hospital length of stay

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as having Veau class II to IV cleft palates undergoing Furlow palatoplasty with ADM between the ages of 3 months and 3 years will be included in this study.

Exclusion Criteria:

* Selection will be based on the parent's willingness to allow their child to participate in the study.
* Children with diagnosed craniofacial syndromes will be excluded from the study due their higher than usual incidence of palatal fistulas.
* Children with known wound healing defects, such as Ehler Danlos syndrome, Pseudoxanthoma Elasticum, will be excluded from the study due to their inherent collagen defects and consequently on the incidence of palatal fistulas.
* Children with Veau class I cleft palates and those who will need/needed any surgical technique other then Furlow palatoplasty will be excluded from the study.

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who present to the Montreal Children's Hospital with a cleft palate (Veau II-IV) that undergo surgical repair between the age of 3 months and 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirko, S Gilardino, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldekhayel SA, Sinno H, Gilardino MS. Acellular dermal matrix in cleft palate repair: an evidence-based review. Plast Reconstr Surg. 2012 Jul;130(1):177-182. doi: 10.1097/PRS.0b013e318254b2dc. PMID 22743882

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Group | Retrospective Group
Started | 65 | 66
Completed | 65 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Group | Retrospective Group | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 59.3 (25) | 66.6 (27.1) | 63 (26.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 32 | 30 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Fistula Formation
Description: Number of patients who developed post palatoplasty fistula
Time Frame: Within 1 year of surgery
Measure: Number; unit: participants
Arm/Group | Prospective Group | Retrospective Group
Number analyzed (Participants) | 65 | 66
participants | 1 | 8

2. Secondary Outcome: Number of Participants With Wound Infection
Description: Number of Participants with Wound Infection post cleft palate repair
Time Frame: Within 1 year of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Group | Retrospective Group
Number analyzed (Participants) | 65 | 66
Participants | 0 | 0

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Prospective Group | Retrospective Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No